CLINICAL TRIAL: NCT06226714
Title: A Randomized, Blinded, Peer-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector) in a Population Aged 18-59 Years
Brief Title: A Clinical Trial of ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197 Vector) in 18-59 Year Olds
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-MCVF-003
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-03

CONDITIONS: Meningococcal Meningitis
Keywords: Vaccine; Peer controlled; Immunogenicity; Safety; 18-59 years
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197) (MCV4) (Experimental): Intramuscular injection, 0.5ml
  Interventions: Biological: MCV4
- ACYW135 Group Meningococcal Polysaccharide Vaccine (MPSV4) (Active Comparator): Subcutaneous iniection, 0.5ml
  Interventions: Biological: MPSV4

INTERVENTIONS:
Biological: MCV4 — 1 dose of MCV4 on Day 0
  Arms: ACYW135 Group Meningococcal Polysaccharide Conjugate Vaccine (CRM197) (MCV4)
Biological: MPSV4 — 1 dose of MSPV4 on Day 0
  Arms: ACYW135 Group Meningococcal Polysaccharide Vaccine (MPSV4)

SUMMARY:
This is a randomized, observer-blind, peer-controlled study. There will be 2 treatment groups, screened subjects were given study numbers in the order of enrollment and randomly assigned to the test and control groups in a 1:1 ratio. Subjects were required to complete a 1-dose immunization program with 0.5 ml of vaccine in both the test and control groups.

ELIGIBILITY:
Inclusion Criteria:

* 18~59 years old at the time of screening.
* Should not have received any meningococcal vaccine in the last 3 years.
* Volunteers have given informed consent, have voluntarily signed an informed consent form, are able and willing to comply with the requirements of the clinical trial protocol, and are able to complete the 180-day study follow-up visit.
* Volunteers have given informed consent, have voluntarily signed an informed consent form, are able and willing to comply with the requirements of the clinical trial protocol, and are able to complete the 180-day study follow-up visit.
* Willingness to discuss medical history with the investigator or physician and to allow access to all medical records relevant to this trial.

Exclusion Criteria:

* Fever before vaccination, axillary temperature >37.0°C.
* History of epilepsy, convulsions or seizures or history or family history of psychiatric disorders.
* Volunteers with current meningitis or a history of meningitis.
* Blood pregnancy-positive or breastfeeding women with a planned pregnancy within 180 days of the volunteer or her partner.
* Hypersensitivity to an ingredient or excipient of the medicinal product used in this clinical trial (mainly: group A meningococcal podophyllotoxin, group C meningococcal podophyllotoxin, group Y meningococcal podophyllotoxin, group W135 meningococcal podophyllotoxin, sucrose, mannitol, sodium chloride, dipotassium hydrogen phosphate trihydrate, potassium dihydrogen phosphate).
* Severe hypertension uncontrolled by medication (at on-site measurement: systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 100 mmHg).
* Previous vaccination-related hospitalizations or emergencies.
* Bleeding constitution or condition associated with prolonged bleeding that investigators consider contraindicated for intramuscular injection.
* Other vaccinations within 14 days.
* Participation in other studies involving interventional studies within 28 days prior to study entry (<28 days) and/or during study participation.
* Other circumstances that, in the judgment of the investigator, make participation in this clinical trial inappropriate.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 840 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Meningococcal antibody positive conversion rates for groups A, C, Y, and W135 in all subjects | 30 days post immunization
Geometric mean titer (GMT) of antibodies to groups A, C, Y, and W135 in all subjects | 30 days post immunization
Incidence of adverse reactions in all subjects | Within 30 mins after immunization
Incidence of adverse reactions/events in all subjects | 7 days post immunization
Incidence of adverse reactions/events in all subjects | Within 30 days after immunization

SECONDARY OUTCOMES:
Meningococcal antibody positivity for groups A, C, Y, and W135 | 30 days post immunization
Geometric mean multiplicity (GMI) of increase for groups A, C, Y, and W135 | 30 days post immunization
Antibody titer ≥1:128 ratio for groups A, C, Y, and W135 | 30 days post immunization
Meningococcal antibody positivity for groups A, C, Y, and W135 in selected subjects | 180 days after immunization
GMT for groups A, C, Y, and W135 in selected subjects | 180 days after immunization
GMI for groups A, C, Y, and W135 in selected subjects | 180 days after immunization
Antibody titer ≥1:128 ratio for groups A, C, Y, and W135 in selected subjects | 180 days after immunization
Incidence of serious adverse events (SAEs) in all subjects | Within 180 days after immunization
Incidence of pregnancy events in all subjects | Within 180 days after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wang, Principal Investigator — Chongqing Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Jiangjin District Center for Disease Control and Prevention, Chongqing
  - Wanzhou District Center for Disease Control and Prevention, Chongqing
  - Yuzhong District Center for Disease Control and Prevention, Chongqing